CLINICAL TRIAL: NCT06186843
Title: Effect of Plant-based Diet on Cardiometabolic and Inflammatory Parameters in Kidney Transplant Recipients
Brief Title: Plant-based Diet for Kidney Transplant Recipients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Muralidharan Jagadeesan, Principal Investigator, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTX-PBD-001
Record Dates: First submitted 2023-10-18; First posted 2024-01-02 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Kidney Disease, Chronic; Transplant Complication; Hypertension; Diabetes Mellitus; Metabolic Syndrome; Inflammation; Kidney Transplant Failure; Dietary Habits
Keywords: Kidney transplant; Lifestyle change; Plant-based diet; Metabolic syndrome; Diabetes; Hypertension; Kidney function; Inflammatory states
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Diabetes Mellitus; Metabolic Syndrome; Inflammation; Feeding Behavior | interventions — Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: A single group of kidney transplant recipients will transition to a plant-based diet and be followed for 24 weeks.
Masking Description: There will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Plant-based diet (Experimental): The group will follow a plant-based diet. Compliance will be checked with dietary questionnaires.
  Interventions: Behavioral: Plant-based diet

INTERVENTIONS:
Behavioral: Plant-based diet — A two week training program will be completed which consists of information, resources and activities that will help participants transition to a plant-based diet. Each day of the program, participants will engage with material that provides information about how a plant-based diet can improve health outcomes, how to cook plant-based meals, what to shop for when eating plant-based, and other information that will help participants become comfortable with this dietary change. In addition, each participant will have a virtual, weekly check-in with one of the investigators. Finally, participants will be encouraged to attend a once monthly group session with all participants.

SUMMARY:
The goal of this clinical trial is to evaluate cardiometabolic and inflammatory parameters in kidney transplant recipients after transitioning to a plant-based diet (PBD). The main aims of the study are as follows:

* To test the feasibility of transiting renal allograft recipients who are > 3 months post-transplant to a PBD
* To study the effect of a PBD on cardiometabolic parameters in kidney transplant recipients
* To assess the effect of a PBD on peripheral blood Th17/Treg ratio and systemic inflammation in kidney transplant recipients

Participants will be asked to:

* Complete a 2-week investigator-designed PBD transition program
* Follow a PBD for a minimum of 16 weeks
* Consent for blood draws, urine samples, and fecal samples along with physical exams
* Complete intermittent food frequency questionnaires and quality of life questionnaires
* Periodically meet with investigators and other study participants

Researchers will compare baseline measurements with future measurements for each participant.

DETAILED DESCRIPTION:
Patients will initially be identified through electronic medical record screening.

Eligible patients will be approached in clinic and informed about the study. Patients who agree to participate will sign the informed consent document to complete enrollment.

Phase 1: Dietary Training (weeks 1-2). Patients receive instruction from a Nephrologist, who is experienced in PBDs and medical student investigators about transitioning to a plant-based diet. Patients will complete a 2 week training program consisting of presentations, videos, informational documents, and group sessions. The program is designed such that at the 2 week point, participants will feel comfortable purchasing, cooking, and eating plant-based foods.

Phase 2: Intervention (weeks 3-18). Patients will consume a PBD under supervision for 16 weeks. Each participant will receive weekly phone calls from the study team and there will be monthly large in-person group sessions.

During Phase 2, there will be an optional, but highly recommended, in person group session that occurs every month. These sessions are designed to facilitate conversations and connections between participants. The sessions will help create a sense of community amongst participants. The group sessions will entail answering participants' questions, having discussions about challenges, and breakout groups will be used so participants can talk in a smaller group environment.

Phase 3: Unsupervised PBD (weeks 19-26). Patients will continue to be followed without dietary supervision.

Dietary compliance will be assessed via food frequency questionnaires (Nutrition Quest) at baseline and weeks 18 and 26. In addition, weekly 1 day food recalls will be collected from participants.

All participants will undergo physical examination at baseline and assessment of interval medical history, medication reconciliation, clinical examination, anthropometric studies (Body mass index (BMI), abdominal circumference and mid-arm circumference) at baseline and weeks 18 and 26 of the study.

Blood, urine, and stool samples will be collected and analyzed at baseline and weeks 10, 18 and 26 of the study.

Two 5 mL vials of blood will be drawn per visit (10 mL) (at baseline, 10, 18, 26 weeks). 40 mL of blood total throughout the study.

Per visit, one 5 mL vial of blood will be used for peripheral blood mononuclear cell (PBMC) prep for flow cytometry. The other 5 mL vial of blood will be used for enzyme-linked immunoassay (ELISA).

30-50 mL of urine will be collected at each visit and processed for urinalysis.

Stool samples will be used to evaluate the composition of the gastrointestinal microbiome.

ELIGIBILITY:
Inclusion Criteria:

* > 3 months post-kidney transplant
* On style immunosuppressive medication
* Without evidence of active infection/ inflammatory conditions
* Estimated glomerular filtration rate > 45ml/min/1.73 m^2
* English speaking
* Reliable internet access

Exclusion Criteria:

* Acute/ chronic allograft rejection
* History of non-compliance
* Advance heart failure
* Liver disease
* Pregnancy
* Malignancy
* Chronic Infection
* Currently following a plant-based diet

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Th17/ Treg ratio | Baseline, week 10, 18, 26
  Th17/Treg cell ratio in peripheral blood. Results expressed as cell frequencies
hsCRP | Baseline, week 10, 18, 26
  Plasma levels measured using enzyme-linked immunosorbent assay (ELISA) expressed as units/ mL
Interleukin (IL) Levels (IL-6, IL-17, IL-21) | Baseline, week 10, 18, 26
  Plasma levels measured using ELISA expressed as units/ mL
Weight | Baseline, week 10, 18, 26
  Kilograms
BMI | Baseline, week 10, 18, 26
  Weight in kilograms (kg) and height (m) in meters will be combined to report BMI kg/m^2
Anthropometry | Baseline, week 18, 26
  Mid arm and abdominal circumference will be measured in centimeters
Blood pressure | Baseline, week 10, 18, 26
  Systolic blood pressure (mmHg)/ Diastolic blood pressure (mmHg)
HbA1c | Baseline, week 10, 18, 26
  mmol/mol and percent (percent of total hemoglobin)
Non-fasting blood glucose | Baseline, week 10, 18, 26
  mg/dL
Total cholesterol | Baseline, week 10, 18, 26
  mg/dL
Food frequency questionnaire | Baseline, week 18, 26
  Nutrient intake and physical activity levels will be calculated
Weekly one day food recall | Once per week at baseline and weeks 3-18
  Dietary compliance will be measured with weekly one day food recall. The percentage of total daily food that is whole food plant-based will be calculated

SECONDARY OUTCOMES:
Estimated glomerular filtration rate | Baseline, week 10, 18, 26
  mL/min/1.73m^2
Creatinine | Baseline, week 10, 18, 26
  mg/dL
Kidney disease and quality of life (KDQOL-36) | Baseline, week 18, 26
  Questions are divided into 5 categories (symptom/problem list; effect of kidney disease; burden of kidney disease; physical health composite; mental health composite). Each category is evaluated on a scale from 0 - 100. Higher scores indicate better outcomes
Changes in gut microbiome | Baseline, week 18, 26
  Stool samples collected at pre-specified time points and analyzed by metagenomics for gut microbiome profile
Low-density lipoprotein (LDL) cholesterol | Baseline, week 10, 18, 26
  mg/dL
High-density lipoprotein (HDL) cholesterol | Baseline, week 10, 18, 26
  mg/dL
Triglycerides | Baseline, week 10, 18, 26
  mg/dL

OTHER OUTCOMES:
Blood electrolytes (Na, K, Cl, Ca, Phosphorous) | Baseline, week 10, 18, 26
  mEq/L
Urine protein | Baseline, week 10, 18, 26
  mg/L
Urine albumin | Baseline, week 10, 18, 26
  mg/L
Urine electrolytes (Na, K, Cl, Ca, Phosphorous) | Baseline, week 10, 18, 26
  mEq/L

CONTACTS AND LOCATIONS:
Overall Officials: Muralidharan Jagadeesan, MD, Principal Investigator — George Washington University
Locations (1):
- Transplant Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
The details of the plan are still being decided.

REFERENCES:
- [Background] Jezior D, Krajewska M, Madziarska K, Kurc-Darak B, Janczak D, Patrzalek D, Boryslawski K, Klinger M. Posttransplant overweight and obesity: myth or reality? Transplant Proc. 2007 Nov;39(9):2772-5. doi: 10.1016/j.transproceed.2007.09.001. PMID 18021984
- [Background] Malgorzewicz S, Woloszyk P, Chamienia A, Jankowska M, Debska-Slizien A. Obesity Risk Factors in Patients After Kidney Transplantation. Transplant Proc. 2018 Jul-Aug;50(6):1786-1789. doi: 10.1016/j.transproceed.2018.02.099. Epub 2018 Mar 13. PMID 29937291
- [Background] Shah B, Newman JD, Woolf K, Ganguzza L, Guo Y, Allen N, Zhong J, Fisher EA, Slater J. Anti-Inflammatory Effects of a Vegan Diet Versus the American Heart Association-Recommended Diet in Coronary Artery Disease Trial. J Am Heart Assoc. 2018 Dec 4;7(23):e011367. doi: 10.1161/JAHA.118.011367. PMID 30571591
- [Background] Tan TG, Sefik E, Geva-Zatorsky N, Kua L, Naskar D, Teng F, Pasman L, Ortiz-Lopez A, Jupp R, Wu HJ, Kasper DL, Benoist C, Mathis D. Identifying species of symbiont bacteria from the human gut that, alone, can induce intestinal Th17 cells in mice. Proc Natl Acad Sci U S A. 2016 Dec 13;113(50):E8141-E8150. doi: 10.1073/pnas.1617460113. Epub 2016 Nov 23. PMID 27911839
- [Background] Raj DS, Sohn MB, Charytan DM, Himmelfarb J, Ikizler TA, Mehrotra R, Ramezani A, Regunathan-Shenk R, Hsu JY, Landis JR, Li H, Kimmel PL, Kliger AS, Dember LM; Hemodialysis Novel Therapies Consortium. The Microbiome and p-Inulin in Hemodialysis: A Feasibility Study. Kidney360. 2021 Jan 15;2(3):445-455. doi: 10.34067/KID.0006132020. eCollection 2021 Mar 25. PMID 35369018
- [Background] Serrano M, Srivastava A, Buck G, Zhu B, Edupuganti L, Adegbulugbe E, Shankaranarayanan D, Kopp JB, Raj DS. Dietary Protein and Fiber Affect Gut Microbiome and Treg/Th17 Commitment in Chronic Kidney Disease Mice. Am J Nephrol. 2022;53(8-9):646-651. doi: 10.1159/000526957. Epub 2022 Nov 7. PMID 36349783
- [Background] Hoogeveen EK, Aalten J, Rothman KJ, Roodnat JI, Mallat MJ, Borm G, Weimar W, Hoitsma AJ, de Fijter JW. Effect of obesity on the outcome of kidney transplantation: a 20-year follow-up. Transplantation. 2011 Apr 27;91(8):869-74. doi: 10.1097/TP.0b013e3182100f3a. PMID 21326138
- [Background] Hill CJ, Courtney AE, Cardwell CR, Maxwell AP, Lucarelli G, Veroux M, Furriel F, Cannon RM, Hoogeveen EK, Doshi M, McCaughan JA. Recipient obesity and outcomes after kidney transplantation: a systematic review and meta-analysis. Nephrol Dial Transplant. 2015 Aug;30(8):1403-11. doi: 10.1093/ndt/gfv214. Epub 2015 Jun 4. PMID 26044837
- [Background] Nicoletto BB, Fonseca NK, Manfro RC, Goncalves LF, Leitao CB, Souza GC. Effects of obesity on kidney transplantation outcomes: a systematic review and meta-analysis. Transplantation. 2014 Jul 27;98(2):167-76. doi: 10.1097/TP.0000000000000028. PMID 24911038
- [Background] Wing MR, Yang W, Teal V, Navaneethan S, Tao K, Ojo A, Guzman NN, Reilly M, Wolman M, Rosas SE, Cuevas M, Fischer M, Lustigova E, Master SR, Xie D, Appleby D, Joffe M, Kusek J, Feldman HI, Raj DS; Chronic Renal Insufficiency Cohort (CRIC) Study. Race modifies the association between adiposity and inflammation in patients with chronic kidney disease: findings from the chronic renal insufficiency cohort study. Obesity (Silver Spring). 2014 May;22(5):1359-66. doi: 10.1002/oby.20692. Epub 2014 Feb 11. PMID 24415732
- [Background] Abedini S, Holme I, Marz W, Weihrauch G, Fellstrom B, Jardine A, Cole E, Maes B, Neumayer HH, Gronhagen-Riska C, Ambuhl P, Holdaas H; ALERT study group. Inflammation in renal transplantation. Clin J Am Soc Nephrol. 2009 Jul;4(7):1246-54. doi: 10.2215/CJN.00930209. Epub 2009 Jun 18. PMID 19541816
- [Background] Nettleton JA, Steffen LM, Palmas W, Burke GL, Jacobs DR Jr. Associations between microalbuminuria and animal foods, plant foods, and dietary patterns in the Multiethnic Study of Atherosclerosis. Am J Clin Nutr. 2008 Jun;87(6):1825-36. doi: 10.1093/ajcn/87.6.1825. PMID 18541574
- [Background] Gutierrez OM, Muntner P, Rizk DV, McClellan WM, Warnock DG, Newby PK, Judd SE. Dietary patterns and risk of death and progression to ESRD in individuals with CKD: a cohort study. Am J Kidney Dis. 2014 Aug;64(2):204-13. doi: 10.1053/j.ajkd.2014.02.013. Epub 2014 Mar 27. PMID 24679894
- [Background] Cyrino LG, Galpern J, Moore L, Borgi L, Riella LV. A Narrative Review of Dietary Approaches for Kidney Transplant Patients. Kidney Int Rep. 2021 Apr 27;6(7):1764-1774. doi: 10.1016/j.ekir.2021.04.009. eCollection 2021 Jul. PMID 34307973
- [Background] Gao B, Alonzo-Palma N, Brooks B, Jose A, Barupal D, Jagadeesan M, Nobakht E, Collins A, Ramezani A, Omar B, Amdur RL, Raj DS. A Pilot Study on the Effect of Prebiotic on Host-Microbial Co-metabolism in Peritoneal Dialysis Patients. Kidney Int Rep. 2020 Jun 1;5(8):1309-1315. doi: 10.1016/j.ekir.2020.05.023. eCollection 2020 Aug. No abstract available. PMID 32775832
- [Background] Amdur RL, Paul R, Barrows ED, Kincaid D, Muralidharan J, Nobakht E, Centron-Vinales P, Siddiqi M, Patel SS, Raj DS. The potassium regulator patiromer affects serum and stool electrolytes in patients receiving hemodialysis. Kidney Int. 2020 Nov;98(5):1331-1340. doi: 10.1016/j.kint.2020.06.042. Epub 2020 Aug 1. PMID 32750456
- [Background] Kalantar-Zadeh K, Kopple JD, Deepak S, Block D, Block G. Food intake characteristics of hemodialysis patients as obtained by food frequency questionnaire. J Ren Nutr. 2002 Jan;12(1):17-31. doi: 10.1053/jren.2002.29598. PMID 11823990
- [Background] Wallace TM, Levy JC, Matthews DR. Use and abuse of HOMA modeling. Diabetes Care. 2004 Jun;27(6):1487-95. doi: 10.2337/diacare.27.6.1487. PMID 15161807